CLINICAL TRIAL: NCT00301483
Title: A Single-Center, Study to Evaluate the Safety and Tolerability of Hemoglobin-Based Oxygen Carrier-201 (HBOC 201) in Trauma Subjects. (Phase II - Safety and Tolerability)
Brief Title: A Single Site Safety and Tolerability Study of HBOC-201 in Trauma Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biopure Corporation (Industry)
Responsible Party: Biopurure Corporation, Biopure
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HEM-0125
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-02

CONDITIONS: Wounds and Injuries
Keywords: multiple trauma; bleeding injuries; gunshot wounds; stab wounds; penetrating injuries; blunt trauma; multiple wounds
MeSH Terms: conditions — Wounds and Injuries; Multiple Trauma; Wounds, Gunshot; Wounds, Stab; Wounds, Nonpenetrating | interventions — HBOC 201; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): HBOC-201 followed by standard therapy
  Interventions: Drug: Hemoglobin-based oxygen carrier-201 (HBOC 201)
- 2 (Active Comparator): Standard Therapy
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Hemoglobin-based oxygen carrier-201 (HBOC 201) — HBOC-201 is an investigational solution of sterile, ultrapurified, glutaraldehyde polymerized, modified bovine hemoglobin (Hb) in a balanced electrolyte solution. HBOC-201 has an Hb concentration of 12-14g/dL. HBOC-201 is an isosmotic solution that is stable for at least 36 months at 2-30ºC. It requires no reconstitution and can be administered directly into a peripheral or central vein. Blood typing is not required because all other cellular components, including the RBC membranes that carry the blood group antigens, have been removed.
  Arms: 1
Other: Standard of Care — Standard Therapy
  Arms: 2

SUMMARY:
The main purpose of this study is to determine if HBOC-201 is safe and tolerable to trauma subjects, when given to treat the inadequate supply of blood and nutrients to tissues and organs.

DETAILED DESCRIPTION:
This Phase II study will be a single-center, randomized, single-blind, parallel-group, standard therapy-controlled, variable dose study of HBOC 201 administered to trauma subjects with bleeding or potential for bleeding who require standard fluid therapy for treatment of hypoperfusion. The type and incidence of adverse events and serious adverse events attributed to the study drug will be analyzed.

Secondary variables in this safety and tolerability study, will be summarized with descriptive statistics and frequency tables. The purpose of this data collection is to assess efficacy variables and the feasibility of utilizing these parameters in future trauma studies that will assess parameters of morbidity and mortality and include, but are not limited to:

* Time to improvement of serum (or plasma) lactate
* Time to improvement in the Base Deficit
* Time to maintained stability (BD<5) over 24 hours
* Overall improvement in Base Deficit over 24 Hours
* Stability of subjects at 24 hours
* Time to meet treatment-stopping criteria
* Volume to meet treatment-stopping criteria
* Incidence of infectious complications (e.g., incidence of ventilator-associated pneumonia)
* Length of time on ventilator
* Incidence of multiple organ dysfunction (MOD)

Hemorrhage with subsequent hypoperfusion is a major cause of both immediate and delayed death in subjects who have sustained traumatic injuries. Effective therapies for hemorrhage to treat hypoperfusion that can be given immediately following injury are lacking. The following issues confound this problem further:

* Hemorrhaging trauma victims often have an immediate need for therapy to ensure adequate delivery of oxygen to vital tissues;
* Standard of care fluids such as Lactated Ringers Solution do not provide oxygen and blood can not be readily stored, transported or easily used in pre-hospital settings
* In the absence of oxygen-carrying fluid, traditional approaches to sustain vital organ perfusion, such as administration of intravenous fluid therapy, may have detrimental effects if given prior to hemostasis in certain subjects, particularly those with penetrating truncal injuries.

ELIGIBILITY:
INCLUSION CRITERIA:

* Male or Female (females not of childbearing potential or negative pregnancy test prior to enrollment)
* Age ≥ 18 years and ≤ 65 years of age
* Trauma with bleeding or a potential for bleeding arriving at initial treatment facility directly from scene of injury
* Subject should be enrolled within four (4) hours of injury
* Base Deficit (BD) greater than 5.0 and one of the following:

Systolic Blood Pressure ≤ 100 mm Hg OR Sustained (≥ 10 minutes) Heart Rate ≥ 100

* No localized signs of traumatic brain injury and a Glasgow Coma Score of ≥9 with the exception of drug-induced lowered GCS.
* Informed consent, or independent physician authorization obtained

EXCLUSION CRITERIA:

* Known or suspected Traumatic Brain Injury
* Non-survivable injury (Falcone Criteria)
* Traumatic arrest
* Known prior cardiac arrest (i.e., preceding trauma episode)
* Known or suspected pregnancy
* Known allergy to bovine products
* Prior treatment with blood (subsequent to current trauma)
* Informed consent or independent physician authorization unable to be obtained
* Unable to meet protocol or follow-up criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2004-07; Primary Completion 2008-09 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Safety/Tolerability of HBOC-201 for treatment of hypoperfusion in trauma by analysis of AEs/SAEs attributed to study drug | Duration of the study (Randomization through 28-day follow-up)

SECONDARY OUTCOMES:
Efficacy/feasibility of the following measurements in trauma studies (list is not all inclusive): Time to serum lactate improvement, Base deficit (BD) improvement, BD > 5 over 24 hrs, 24 hr stability, Infection, Vent time | Duration of the study (Randomization through 28-day follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: A. Gerson Greenburg, MD, PhD, Study Director — Biopure Corporation; Professor Ken D Boffard, MD, Principal Investigator — Wits University Medical School
Locations (1):
- Department of Surgery: Johannesburg Hospital, Johannesburg, Gauteng, South Africa